CLINICAL TRIAL: NCT01116908
Title: Safe Drinking Water For Households With Infants Born to HIV-Positive Mothers in Zambia: Piloting a Household Water Treatment Intervention
Brief Title: Safe Drinking Water For Households With Infants Born to HIV-Positive Mothers Pilot Study
Acronym: SWIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other); University of Zambia (Other); Vestergaard Frandsen (Other)
Responsible Party: Dr. Thomas Clasen, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QA270
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Diarrhea; HIV Infection
Keywords: Diarrhea; Water; Household Water Treatment; HIV; Infant Health
MeSH Terms: conditions — Diarrhea; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- LifeStraw Family (Active Comparator)
  Interventions: Device: LifeStraw Family

INTERVENTIONS:
Device: LifeStraw Family — LifeStraw Family is a household water treatment technology that will be implemented in the household to improve drinking water quality
  Arms: LifeStraw Family

SUMMARY:
The purpose of this study is to assess whether children under 2 years and other members of households in which HIV-positive mothers are providing replacement and complementary feeding would potentially benefit from the use of a filter designed to eliminate microbial pathogens from drinking water at the household level.

DETAILED DESCRIPTION:
Contaminated drinking water is a leading cause of morbidity and mortality in low-income settings. Safe drinking water is of particular concern for HIV-positive mothers since many HIV-infected Zambian women choose replacement feeding and early cessation of breastfeeding of infants to minimize the risk of transmission of the virus. This study builds upon preliminary baseline research which determined that HIV-positive mothers would potentially benefit from an intervention that encourages HIV-positive mothers to treat their water at the household level.

ELIGIBILITY:
Inclusion Criteria:

* Known HIV-status based on clinical testing
* Have a child between 6-12 months at the initiation of the study
* Within the catchment area of Kasisi or Ngwerere health clinics, Chongwe district, Lusaka

Exclusion Criteria:

* Lived in the catchment area less than one year or planning to move

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Use of LifeStraw Family for children under 2 and all household members | One year
  Use, acceptability, and longevity of LifeStraw Family will be assessed for replacement and complementary feeds for children under 2 and for drinking water for all members of the household

SECONDARY OUTCOMES:
Microbiological performance of LifeStraw Family | One year
  Microbiological performance of LifeStraw Family, measured in terms of thermotolerant coliforms (TTC), a well-established WHO indicator organism for faecal contamination
Impact of LifeStraw Family on longitudinal prevalence of diarrhea | One year
  Impact of the intervention on longitudinal prevalence of diarrhoea among infants under 2 years and all household members, measured both as reported by the primary caretaker of the child and by their weight-for-age z-score (WAZ) as a proxy for diarrhoea

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Clasen, JD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Ngwerere Health Clinic and Kasisi Health Clinic, Lusaka, Chongwe District, Lusaka Province, Zambia

REFERENCES:
- [Derived] Peletz R, Simunyama M, Sarenje K, Baisley K, Filteau S, Kelly P, Clasen T. Assessing water filtration and safe storage in households with young children of HIV-positive mothers: a randomized, controlled trial in Zambia. PLoS One. 2012;7(10):e46548. doi: 10.1371/journal.pone.0046548. Epub 2012 Oct 17. PMID 23082124